CLINICAL TRIAL: NCT04892628
Title: Measurement of Subjective and Objective Indices After Progressive Resistance Training Compared With Aerobic Training in Patients With Hemophilia: a Randomised Controlled Trial
Brief Title: Effects of Progressive Resistance Training Compared With Aerobic Training in Patients With Hemophilia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Felicianus Pereira, Principal Investigator - Postgraduate Trainee, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Hem_resistance_aerobic_pk
Record Dates: First submitted 2021-05-04; First posted 2021-05-19 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Quality of Life; Muscle Weakness
Keywords: Hemophilia; resistance training; aerobic exercise; Pakistan
MeSH Terms: conditions — Muscle Weakness; Hemophilia A

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic training group (Other): The control group will be administered a standard physical therapy intervention program which will consist of active muscle stretching and aerobic exercises.
  Exercises will include:
  * Flexion, extension and abduction at the shoulder joint for anterior, middle and posterior fibers of deltoid
  * Flexion and extension at the elbow for biceps and triceps trachii
  * Flexion and extension at the knee joint for quadriceps and hamstring muscles
  * Plantar flexion at the ankle joint for gastrocnemius and soleus
  Three sets of ten repetitions of each exercise will be done.
  Interventions: Other: Aerobic training
- Resistance training group (Experimental): The intervention group will undergo a progressive resistance training program consisting of active muscle stretching and resistance training. Exercise for intervention group will consist of:
  * Resisted flexion, extension and abduction at the shoulder joint for anterior, middle and posterior deltoid, using dumbbells
  * Resisted flexion and extension at the elbow for biceps and triceps trachii, using dumbbells
  * Resisted flexion and extension of knee joint for quadriceps and hamstring muscles, using therabands
  * Resisted dorsiflexion and plantar flexion of gastrocnemius and soleus, using therabands
  Resistance will be increased on basis of progressive overload principle. Three sets of ten repetitions will be performed per muscle group. Initial weight of the dumbbells will be 1kg and will be increased by 0.5kg per week.
  Interventions: Other: Progressive resistance training

INTERVENTIONS:
Other: Progressive resistance training — Resistance training of upper limb and lower limb muscles. Resistance will be increased on a weekly basis. Dumbbells and therabands will be used to provide resistance.
  Arms: Resistance training group
Other: Aerobic training — The control group will be administered a standard physical therapy intervention program which will consist of active muscle stretching and aerobic exercises.
  Arms: Aerobic training group

SUMMARY:
This study aims to assess the effects of progressive resistance training compared with aerobic training, among those with hemophilia. Participants will be divided into two groups. The control group will receive an aerobic exercise protocol, and the resistance group will follow a resistance training program. Each group will receive a total of eight sessions. Target muscles are deltoids, biceps, triceps, quadriceps, hamstrings, and calves.

Subjective and objective assessment will be performed for each group, to determine the effectiveness of each intervention.

DETAILED DESCRIPTION:
Participant's height, weight and age will be recorded for pre-test anthropometric data. Height will be measured using a stadiometer, and weight will be measured with an electronic scale.

Treatment sessions will be conducted twice a week, for 8 weeks. The control group will be administered a standard physical therapy intervention program which will consist of active muscle stretching and aerobic exercises.

Exercises will include:

* Flexion, extension and abduction at the shoulder joint for anterior, middle and posterior fibers of deltoid
* Flexion and extension at the elbow for biceps and triceps trachii
* Flexion and extension at the knee joint for quadriceps and hamstring muscles
* Plantar flexion at the ankle joint for gastrocnemius and soleus Three sets of ten repetitions of each exercise will be done.

The intervention group will undergo a progressive resistance training program consisting of active muscle stretching and resistance training. Exercise for intervention group will consist of:

* Resisted flexion, extension and abduction at the shoulder joint for anterior, middle and posterior deltoid, using dumbbells
* Resisted flexion and extension at the elbow for biceps and triceps trachii, using dumbbells
* Resisted flexion and extension of knee joint for quadriceps and hamstring muscles, using therabands
* Resisted dorsiflexion and plantar flexion of gastrocnemius and soleus, using therabands

Resistance will be increased on basis of progressive overload principle. Three sets of ten repetitions will be performed per muscle group. Initial weight of the dumbbells will be 1kg and will be increased by 0.5kg per week. Therabands used will be Yellow, Red, Green and Blue. Resistance for therabands will be upgraded every two weeks. Treatment time per group will be approximately 40 minutes. Exercises will be progressed in a gradual manner to give participants time to build muscle strength.

ELIGIBILITY:
Inclusion Criteria:

* clinically diagnosed with hemophilia A or B (mild to moderate hemophilia (mild hemophilia - 0.05-0.4 IU, moderate hemophilia - 0.01-0.05 IU)
* undergo pre- and post-program objective assessment of manual muscle testing and Hemophilia Joint Health Score, as well as subjective assessment of and Rating of Perceived Exertion.
* willing to train two times a week
* males and females between 18 to 45 years of age.
* those who can ambulate without assistance

Exclusion Criteria:

* unable to attend exercise sessions for the complete duration of the study
* those who have had surgery performed 6 weeks before, or in duration of training (due to any disability)
* involvement in any other training, or rehabilitation, during study
* change in medicine within the study
* history of major bleeding episodes that could pose a risk
* history of factor 8 or factor 9 inhibitor

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-04-03 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Manual Muscle Testing - Daniel & Worthingham's | baseline and post intervention (week 8 - the analysis will be conducted on the first week immediately after the end of the training)
  An objective marker to determine muscle strength. It ranges from 0-5
  0 no movement of muscle
  1. flickering movement of muscle
  2. full range of motion in a gravity minimized position
  3. full range of motion against gravity, without resistance
  4. muscle can hold against moderate resistance
  5. muscle can hold against maximal resistance
Hemophilia Joint Health Score (HJHS v2.1) | baseline and post intervention (week 8 - the analysis will be conducted on the first week immediately after the end of the training)
  The HJHS measures joint health, in the domain of body structure and function (i.e. impairment), of the joints most commonly affected by bleeding in hemophilia: the knees, ankles, and elbows. It can be used when there is a need for orthopedic intervention, or as an outcome measure of physiotherapy interventions.
  A scoring system is present, which combines the score of these questions, with a global gait score, to give an overall score. The greater the score, the poorer the outcome.
  The HJHS 2.1 provides a total score (higher score is worse; max=124), joint specific scores, and a global gait score.
Borg Rating of Perceived Exertion | baseline and post intervention (week 8 - the analysis will be conducted on the first week immediately after the end of the training)
  The second subjective marker. This will be used to assess the subjective workload of exercises, and to note if exercise intensity decreases over time.
  The values range from 6-20, with 6 rated as 'no exertion', and 20 rated as 'maximal exertion'.
HEP-Test-Q (Hemophilia and Exercise Project) | baseline and post intervention (week 8 - the analysis will be conducted on the first week immediately after the end of the training)
  The subjective marker of this study. This measure will assess the quality of life. It is a scale specifically designed for people with hemophilia.
  The HEP-Test-Q consists of 25 items pertaining to 4 domains 'mobility', 'strength & coordination', 'endurance' and 'body perception' and one single item, which assesses changes in physical functioning in comparison to the previous year.
  The recall period for the assessment of physical functioning is over "the past four weeks".
  The response options range on a 5-point Likert scale from "never" to "always".
  Some of the items have to be re-coded. Subscales and the total score are transformed to a scale of 0-100 with high scores indicating better physical functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Pereira, Principal Investigator — Dow University of Health Sciences
Locations (1):
- Hemophilia welfare society karachi, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Parhampour B, Dadgoo M, Vasaghi-Gharamaleki B, Torkaman G, Ravanbod R, Mirzaii-Dizgah I, Reza Baghaipour M, Saneii SH. The effects of six-week resistance, aerobic and combined exercises on the pro-inflammatory and anti-inflammatory markers in overweight patients with moderate haemophilia A: A randomized controlled trial. Haemophilia. 2019 Jul;25(4):e257-e266. doi: 10.1111/hae.13764. Epub 2019 May 26. PMID 31131517